CLINICAL TRIAL: NCT06483906
Title: Efficacy and Safety of Venetoclax and Azacitidine Combined With Low-Intensity Homoharringtonine Chemotherapy Followed by Allogeneic Hematopoietic Stem Cell Transplantation in Intermediate/High-Risk Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Venetoclax and Azacitidine Combined With Homoharringtonine, Followed by Allo-HSCT for Intermediate and High-risk AML.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-202403-VAH
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; allogeneic hematopoietic stem cell transplantation; Venetoclax; Azacitidine; Homoharringtonine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VAH regimen combined with allo-HSCT (Experimental): Eligible patients receive two cycles of the VAH chemotherapy regimen. If minimal residual disease (MRD) is negative after these two cycles, patients proceed to the transplantation process. If MRD remains positive, patients receive an additional two cycles of the VAH regimen. Upon achieving MRD negativity, they then proceed to the transplantation process.
  Interventions: Drug: Venetoclax, Azacitidine and Homoharringtonine

INTERVENTIONS:
Drug: Venetoclax, Azacitidine and Homoharringtonine — Patients will receive the VAH regimen for the treatment of AML
  Other Names: VAH

SUMMARY:
This study is a single-center, single-arm, prospective phase II clinical trial evaluating the efficacy and safety of the VAH (Venetoclax and Azacitidine combined with Homoharringtonine) regimen, followed by allo-HSCT for intermediate and high-risk AML. Eligible patients receive two cycles of the VAH chemotherapy regimen. If minimal residual disease (MRD) is negative after these two cycles, patients proceed to the transplantation process. If MRD remains positive, patients receive an additional two cycles of the VAH regimen. Upon achieving MRD negativity, they then proceed to the transplantation process.

The conditioning regimen includes fludarabine at 30 mg/m²/day from day -7 to day -3 (5 days), cytarabine at 1-1.5 g/m²/day from day -7 to day -3 (5 days), and busulfan at 3.2 mg/kg/day from day -5 to day -3 (3 days). Conditioning begins on day -6, and donor hematopoietic stem cell infusion is performed on day 0.

All patients will undergo bone marrow examination on day 14 and day 28 post-transplant, followed by bone marrow examinations every 30 days within the first year after transplantation, and every 60 days within the second year. If disease relapse is suspected during the follow-up period, bone marrow or extramedullary relapse site examinations will be conducted at any time.

The primary endpoint is the 1-year and 2-year overall survival (OS). Secondary endpoints include the complete response (CR) rate after 1 and 2 cycles of chemotherapy; 1-year and 2-year disease-free survival (DFS) following the achievement of CR through induction therapy; cumulative relapse rate; non-relapse mortality (NRM); incidence of acute graft-versus-host disease (GVHD) within 180 days post-transplant; and the cumulative incidence of chronic GVHD within 1 year and 2 years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 55 years, inclusive, regardless of gender.
2. Diagnosed with AML (excluding APL) according to the 2022 International Consensus Classification (ICC) for AML [1].
3. Evaluated as intermediate/high-risk AML based on the 2022 ELN AML guidelines (see Appendix 1).
4. No prior treatment for acute leukemia, including hypomethylating agents used for leukemia or myelodysplastic syndromes (MDS), except for hydroxyurea.
5. Patients must have a suitable hematopoietic stem cell donor.
6. Hematopoietic cell transplantation comorbidity index (HCT-CI) score ≤ 2.
7. ECOG (Eastern Cooperative Oncology Group) performance status: 0-2.
8. Adequate liver, kidney, and cardiopulmonary function, meeting the following requirements:

   1. Serum creatinine ≤ 1.5x ULN (the upper limit of normal);
   2. Cardiac function: Ejection fraction ≥ 50%;
   3. Baseline oxygen saturation > 92%;
   4. Total bilirubin ≤ 1.5 x ULN; ALT and AST ≤ 2.0 x ULN;
   5. Pulmonary function: DLCO (corrected for hemoglobin) ≥ 40% and FEV1 (Forced Expiratory Volume in 1 second) ≥ 50%.

      9) Patients must have the ability to understand and be willing to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Presence of extramedullary disease manifestations at diagnosis or during treatment, including central nervous system involvement.
3. History of malignancies other than myeloid neoplasms within the past 5 years prior to screening, except adequately treated cervical carcinoma in situ, basal cell carcinoma, squamous cell carcinoma of the skin, and localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery.

4) ECOG > 2. 5) HCT-CI score ≥ 3. 6) Any unstable systemic diseases, including but not limited to unstable angina, recent cerebrovascular accidents or transient ischemic attacks within the 3 months prior to screening, myocardial infarction within the 3 months prior to screening, congestive heart failure (New York Heart Association [NYHA] class ≥ III), severe arrhythmias requiring drug treatment after pacemaker implantation, significant liver, kidney, or metabolic diseases, and pulmonary arterial hypertension.

7) Active, uncontrolled infections, including those associated with hemodynamic instability, new or worsening infection symptoms or signs, new infectious lesions on imaging, or persistent unexplained fever without signs or symptoms of infection.

8) Conditions requiring treatment such as grade 2 or higher seizures, paralysis, aphasia, recent severe cerebral infarction, severe traumatic brain injury, dementia, Parkinson's disease, or schizophrenia.

9) HIV-infected individuals. 10) Active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral therapy.

Patients at risk of HBV reactivation, are defined as those who are positive for hepatitis B surface antigen or core antibody without receiving antiviral therapy.

11) History of autoimmune diseases. 12) Pregnant or breastfeeding women. 13)Fertile males and females unwilling to use contraception during the treatment period and for 12 months after treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
1y and 2y-OS | up to 2 years
  1-year and 2-year overall survival (OS) after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arber DA, Orazi A, Hasserjian RP, Borowitz MJ, Calvo KR, Kvasnicka HM, Wang SA, Bagg A, Barbui T, Branford S, Bueso-Ramos CE, Cortes JE, Dal Cin P, DiNardo CD, Dombret H, Duncavage EJ, Ebert BL, Estey EH, Facchetti F, Foucar K, Gangat N, Gianelli U, Godley LA, Gokbuget N, Gotlib J, Hellstrom-Lindberg E, Hobbs GS, Hoffman R, Jabbour EJ, Kiladjian JJ, Larson RA, Le Beau MM, Loh ML, Lowenberg B, Macintyre E, Malcovati L, Mullighan CG, Niemeyer C, Odenike OM, Ogawa S, Orfao A, Papaemmanuil E, Passamonti F, Porkka K, Pui CH, Radich JP, Reiter A, Rozman M, Rudelius M, Savona MR, Schiffer CA, Schmitt-Graeff A, Shimamura A, Sierra J, Stock WA, Stone RM, Tallman MS, Thiele J, Tien HF, Tzankov A, Vannucchi AM, Vyas P, Wei AH, Weinberg OK, Wierzbowska A, Cazzola M, Dohner H, Tefferi A. International Consensus Classification of Myeloid Neoplasms and Acute Leukemias: integrating morphologic, clinical, and genomic data. Blood. 2022 Sep 15;140(11):1200-1228. doi: 10.1182/blood.2022015850. PMID 35767897
- [Background] Kantarjian HM, Kadia TM, DiNardo CD, Welch MA, Ravandi F. Acute myeloid leukemia: Treatment and research outlook for 2021 and the MD Anderson approach. Cancer. 2021 Apr 15;127(8):1186-1207. doi: 10.1002/cncr.33477. Epub 2021 Mar 18. PMID 33734442
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] De Kouchkovsky I, Abdul-Hay M. 'Acute myeloid leukemia: a comprehensive review and 2016 update'. Blood Cancer J. 2016 Jul 1;6(7):e441. doi: 10.1038/bcj.2016.50. PMID 27367478
- [Background] Fernandez HF, Sun Z, Yao X, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald GW, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Tallman MS. Anthracycline dose intensification in acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1249-59. doi: 10.1056/NEJMoa0904544. PMID 19776406
- [Background] Lee JH, Joo YD, Kim H, Bae SH, Kim MK, Zang DY, Lee JL, Lee GW, Lee JH, Park JH, Kim DY, Lee WS, Ryoo HM, Hyun MS, Kim HJ, Min YJ, Jang YE, Lee KH; Cooperative Study Group A for Hematology. A randomized trial comparing standard versus high-dose daunorubicin induction in patients with acute myeloid leukemia. Blood. 2011 Oct 6;118(14):3832-41. doi: 10.1182/blood-2011-06-361410. Epub 2011 Aug 9. PMID 21828126
- [Background] Percival ME, Tao L, Medeiros BC, Clarke CA. Improvements in the early death rate among 9380 patients with acute myeloid leukemia after initial therapy: A SEER database analysis. Cancer. 2015 Jun 15;121(12):2004-12. doi: 10.1002/cncr.29319. Epub 2015 Mar 4. PMID 25739348
- [Background] Mi R, Zhao J, Chen L, Wei X, Liu J, Wei X. Efficacy and Safety of Homoharringtonine for the Treatment of Acute Myeloid Leukemia: A Meta-analysis. Clin Lymphoma Myeloma Leuk. 2021 Oct;21(10):e752-e767. doi: 10.1016/j.clml.2021.06.002. Epub 2021 Jun 9. PMID 34301487
- [Background] Tang R, Faussat AM, Majdak P, Marzac C, Dubrulle S, Marjanovic Z, Legrand O, Marie JP. Semisynthetic homoharringtonine induces apoptosis via inhibition of protein synthesis and triggers rapid myeloid cell leukemia-1 down-regulation in myeloid leukemia cells. Mol Cancer Ther. 2006 Mar;5(3):723-31. doi: 10.1158/1535-7163.MCT-05-0164. PMID 16546987
- [Background] Shi Y, Ye J, Yang Y, Zhao Y, Shen H, Ye X, Xie W. The Basic Research of the Combinatorial Therapy of ABT-199 and Homoharringtonine on Acute Myeloid Leukemia. Front Oncol. 2021 Jul 14;11:692497. doi: 10.3389/fonc.2021.692497. eCollection 2021. PMID 34336680
- [Background] Jin H, Zhang Y, Yu S, Du X, Xu N, Shao R, Lin D, Chen Y, Xiao J, Sun Z, Deng L, Liang X, Zhang H, Guo Z, Dai M, Shi P, Huang F, Fan Z, Yin Z, Xuan L, Lin R, Jiang X, Yu G, Liu Q. Venetoclax Combined with Azacitidine and Homoharringtonine in Relapsed/Refractory AML: A Multicenter, Phase 2 Trial. J Hematol Oncol. 2023 Apr 29;16(1):42. doi: 10.1186/s13045-023-01437-1. PMID 37120593